CLINICAL TRIAL: NCT03152110
Title: Feasibility and Acceptability of Six-weeks of High Intensity Interval Training in Wheelchair Users With SCI
Brief Title: Feasibility of HIIT in Spinal Cord Injury
Acronym: HIIT-SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Alabama at Birmingham (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alicia Koontz, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO17020277; 1P2CHD086851 (NIH)
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: High Intensity Interval Training; HIIT; Physical Activity
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIIT (Experimental): Exercise sessions will be 3x/week for 6 weeks (2 sessions supervised, 1 session unsupervised). The HIIT goal is to achieve 10 sets of 60 second bouts of arm cycling at 90% of their PPO with 60 seconds of active recovery.
  Interventions: Other: HIIT

INTERVENTIONS:
Other: HIIT — A handcycle or tabletop ergometer will be used for HIIT. Exercise sessions will be scheduled 3x/week for 6 weeks (2 sessions supervised, 1 session unsupervised). The HIIT goal is to achieve 10 sets of 60 second bouts of arm cycling at 90% of their PPO with 60 seconds of active recovery.
  Supervised exercise sessions: Measures include HR, BP, RPEs, Feeling Scale, and PPO. After warming up, individualized work/rest phases will be prescribed based on their PPO from their maximal aerobic test. Participants will be held at 90% PPO as a constant target intensity to start, shortening the work phase, and if necessary, lengthening the recovery phase. These parameters will be progressed each session. The trainer will determine when to change their work/rest parameters based off of HR and RPEs.
  Unsupervised exercise sessions: Participants will repeat the same HIIT protocol they performed during the previous supervised session. The bike computer automatically stores HR and PPO.

SUMMARY:
Spinal cord injury (SCI) is debilitating to an individual's health, functional capacity and quality of life. This contributes to a sedentary lifestyle and an elevated risk for cardiometabolic and hypokinetic diseases. While physical activity is promoted in persons with SCI to reduce incidence of secondary disabling conditions, a majority of individuals are inactive and have low levels of fitness. High intensity interval training (HIIT) is a form of exercise characterized by brief, intermittent bouts of intense exercise, separated by periods of lower intensity exercise for recovery. The level of improvements in aerobic exercise capacity following HIIT are similar to moderate-intensity continuous training, but only require a fraction of the total energy and time commitment. Little research has been done on HIIT in persons with SCI, who are unable to carry out conventional lower limb HIIT exercises. An upper extremity form of HIIT that is effective, safe, and quick could be an attractive option for these individuals. The study will look at feasibility and acceptability of a 6-week HIIT program for persons with a spinal cord injury who are untrained.

Investigators will test 10 untrained individuals with SCI/D who use a manual wheelchair full time. Prior to any testing, participants will be screened and will need to obtain a signed medical release from their physician. The screening involves asking the participant the inclusion/exclusion criteria and administering two short questionnaires related to physical activity. After obtaining the release form, participants will be scheduled for their first visit. During Visit 1, baseline testing and questionnaires will be completed. The study questionnaires will address sociodemographics, pain and health measures, general health, and physical activity. Exercise testing includes an aerobic exercise stress test (conducted following American College of Sports Medicine guidelines using an electronic ergometer) and an anaerobic (maximum power output) test. After Visit 1, participants will exercise three times per week for six weeks, following a standard HIIT protocol. Two of those sessions will be supervised by a trainer, and one session will be completed on their own. After six weeks, participants will be scheduled for Visit 2 and will complete the same evaluations as Visit 1. Additionally, participants will complete evaluations on their level of satisfaction of the training program and their likelihood to continue.

DETAILED DESCRIPTION:
Eligible participants will be sent a physician release form to be signed prior to study initiation. Upon receipt, the participant will be scheduled for their Visit 1, Baseline Visit and will be given the following instructions:

Do not participate in any strenuous physical activity 24 hours prior to testing.

Do not eat a large meal 4 hours prior to testing, however a light snack is okay.

Do not drink alcohol or caffeine 4 hours prior to testing. No smoking 1 hour prior to testing. Wear comfortable, loose clothing that is easy to exercise in.

Visit 1: Baseline Visit

After written informed consent has been obtained, participants will be asked to complete study questionnaires and perform baseline exercise tests. Participants will be asked complete the following questionnaires:

Demographics questionnaire: May include information such as disability type, level of SCI, years with disability, age, gender, and information about their wheelchair.

Numerical Rating Scale (NRS): Participants will complete this scale once for each upper limb joint (wrist, elbow and shoulder). Participants will be asked to rate their average, most severe, and least severe wrist, elbow and shoulder pain during the last 24 hours using an 11 point scale (i.e. 0-10) anchored at the ends by "no pain" and "worst pain ever experienced." An 11-point NRS measure of intensity allows for comparison across clinical trials of pain treatment and is recommended as a core outcome measure for chronic pain clinical trials. NRS pain measures are widely used and have been shown to be valid and reliable assessments of pain.

Wheelchair Users Shoulder Pain Index (WUSPI): This is a 15 item, self-report instrument that measures shoulder pain intensity, within the last week, in wheelchair users during various functional daily activities such as transfers, leading a wheelchair into a car, wheelchair mobility, dressing, bathing, overhead lifting, driving, performing household chores and sleeping. The WUSPI is a valid and reliable measure of shoulder pain. Test-retest reliability of the total index score was 0.99 and Cronbach's alpha (internal consistency) was 0.98.

Short Form Health Survey Walk Wheel (SF-36 WW): A 36-item general health and function questionnaire that has been validated for persons with SCI. The SF-36 is a brief, multi-dimensional, self-report health questionnaire that measures eight concepts: physical functioning, role limitation due to physical problems, bodily pain, general perception of health, vitality, social function, role limitation due to emotional problems and mental health.

Physical Activity Scale for Individuals with Physical Disabilities (PASIPD): The PASIPD is a 13-item self-report instrument covering (1) leisure activities, (2) household activities, (3) occupational activities and (4) light, moderate, and strenuous sport and recreational activities. The scale asks individuals to report how many days and hours per week that they spend participating in these various physical activities and a total score is calculated that is expressed in a metabolic equivalent (MET). The maximum possible score on the PASIPD total score is 199.5 MET.

Height and weight will be taken. Subjects will transfer to a mat table where they will lay on their backs. In this position, we will measure their height with a measuring tape. Weight will be calculated using a wheelchair scale as the difference between the weight of the participant in their wheelchair and the weight of the wheelchair alone.

Following completion of all study questionnaires, participants will begin exercise testing administered by an exercise physiologist and directly supervised by a physician. The tests are outlined in further detail below:

Maximal aerobic exercise test: the purpose of this test is to evaluate cardiac function and fitness and determine peak power output (PPO). PPO will later be used to set an individualized goal for the HIIT protocol. Prior to starting the maximal exercise testing, participants will be fitted with a mask that analyzes the inhaled and exhaled air (also known as "open circuit spirometry"). Cardiorespiratory measures (i.e., heart rate, blood pressure, oxygen consumption, respiratory exchange ratio, pulmonary ventilation, carbon dioxide expiration, etc.) will be recorded throughout this test. Heart rate will be collected using the same heart rate monitor that will be worn during the in-home exercise portion of the study. The heart rate monitors will be worn around the chest in area under the heart. Participants will be able to use a private space to put the heart rate monitor on prior to staring the study. A member of the study team will verify the heart rate monitor is placed properly. Prior to beginning the maximal exercise test, the Borg and Wheel Rating of Perceived Exertion (RPE) scales will be presented to participants. RPE scales rate how hard a person feels their body is working and is an accepted supplementary tool for prescribing exercise programs in both healthy and special populations. Throughout the test, the participant will be asked to report their RPE by pointing to the corresponding number on the scales. The exercise test will be administered using an incremental modified Bruce protocol on an electronically braked cycle ergometer. The Bruce protocol outlines speeds and inclines to test cardiopulmonary function and health. The protocol outlines specific time increments and the settings for the treadmill to ensure a maximal aerobic capacity is achieved. This protocol will be modified for an arm ergometer, where the resistance on the ergometer and the revolutions per minute (RPMs) will be modified instead of incline and speed. The settings on the ergometer will attempt to match the incremental changes outlined in the Bruce protocol. Initially, resistance will be set at 25W, and then increased by 25W every 2 minutes until the subject can no longer continue or until their respiratory exchange ratio exceeds 1.15.

Maximum power output test: the primary purpose of this test is to evaluate the highest amount of power that the participant can produce in a short period of time. Other measures include heart rate, blood pressure, relative peak power, anaerobic capacity and anaerobic fatigue. This test will use the same ergometer as the maximal aerobic exercise test. Initially, the resistance will be set at zero and increased over the duration of the test. The participant will initially crank on the cycle with minimal resistance for about thirty seconds, then the resistance will be increased to a maximal level. Participants will crank for as long and as hard as they are able to for another thirty seconds. The participant will be asked to complete this process up to three separate times, with a minimum of 30 seconds of rest in between. After the test is completed, the resistance will return to zero and the participants will cycle at a comfortable pace to cool down.

Following completion of the exercise tests, the study team will introduce the participant to the type of exercises that will be performed for the study. They will be able to use the ergometer in the lab to try out a brief HIIT protocol.

6-Week HIIT Protocol: If the participant owns a handcycle, investigators will attempt to fit their handcycle to the roller system. The study team will provide a handcycle those that do not fit the roller system or individuals who do not own one. If a participant is uncomfortable using a handcycle, or is unable to transfer into the handcycle, the study team will provide a tabletop ergometer. At the end of the study the handcycle or tabletop ergometer and the roller system will be returned to the study team. Participants will be given a heart rate monitor, which they will be asked to wear and use for every exercise session for the duration of the study. They do not have to return the heart rate monitor at the end of the study. Participants will be provided with a bike computer that will be fit to the handcycle/ergometer and will be used for recording power output and heart rate during the exercise sessions. Participants must return the bike computer at the end of the study.

The first exercise visit will be scheduled within one week of the first study visit. Exercise sessions will be scheduled 3 times per week (every other weekday), with the total training protocol lasting 6 weeks. Two of the sessions will be supervised by a trainer and one session will be completed on their own. During the last week (week 6), subjects can opt to have their supervised sessions via FaceTime or Skype (if they have a smartphone or computer). The participant exercise goal is to achieve 10 sets of 60 second bouts of arm cycling at 90% of their PPO (as determined in baseline testing), separated by 60 seconds of active recovery.

(A) Supervised exercise sessions: the trainer will meet the participant at their home for each supervised exercise session. Prior to exercise, the trainer will measure/record the participant's heart rate and blood pressure. In addition, the trainer will make sure that there haven't been any recent changes in health or medical status.

The trainer will guide the participant through a warm-up and stretching routine prior to exercising (approximately 10 minutes). The participant will be familiarized with the same Borg and Wheel RPE scales used during Visit 1, and the Feeling Scale. The Feeling Scale (-5 very bad to +5 very good) is commonly used to measure affective response during exercise.

The trainer will prescribe individualized work and rest phases based on their maximal aerobic test PPO. To reach their HIIT goal, trainers will hold participants at 90% PPO as a constant target intensity to start, shortening the work phase (e.g. 10-15 seconds), and if necessary, lengthening the recovery phase (e.g. 75-90 seconds). These ramping parameters will be progressed and documented by the trainer for each session. The trainer will determine when to change their work and rest parameters based off heart rate and self-reported RPE.

At the end of each session, the trainer will measure/record the participant's heart rate and blood pressure again. Power output and heart rate data is automatically stored in the bike computer during each exercise session to track adherence to the prescribed HIIT intensities.

(B) Unsupervised exercise sessions: participants will be asked to repeat the same HIIT protocol they performed during the previous supervised session. The trainer will provide written directions. Participants will be instructed to wear the heart rate monitor so that during the next supervised exercise session, the trainer will be able to retrieve/collect the data to store on one of our study devices for future analysis. The heart rate data as well as power output data will automatically be stored on the device in the same manner as during the supervised sessions. At the next supervised session the trainer will retrieve the data from the device.

Visit 2:

After completing the 6-week HIIT program, participants will be scheduled for a second/final lab visit. Visit 2 will be scheduled within one week or up to two weeks after finishing the 6-week HIIT program, but to provide scheduling flexibility, participants have up to two weeks to complete their second visit. Investigators will try to schedule the follow-up exercise testing around the same time of day as Visit 1. Participants will complete the same exercise testing protocol that was completed in Visit 1. Participants will also complete the NRS, WUSPI, and SF-36 WW questionnaires from Visit 1and will be asked to complete a survey regarding their satisfaction with the program using the Physical Activity Enjoyment Scale (PACES). Finally, participants will be provided with an open-ended questionnaire to discuss their feelings about HIIT, likelihood to continue, and support needs to help them (or others like them) keep doing HIIT.

ELIGIBILITY:
Inclusion Criteria:

1. SCI/D which occurred at least 6 months prior to the start of the study
2. uses a manual wheelchair as primary means of mobility (30+ hours per week)
3. is between 18 and 65 years of age
4. Weighs less than 250lbs
5. lives within one hour driving time from the research center
6. is able to perform a transfer independently to and from a wheelchair
7. has adequate strength and upper extremity function to operate a handcycle or arm ergometer
8. has adequate space in a safe location (i.e., home, work) to accommodate a handcycle or tabletop ergometer
9. Receipt of a signed physicians medical release form

Exclusion Criteria:

1. History of fractures or dislocations in the upper extremity from which the participant has not fully recovered
2. Upper limb pain or injury that interferes with the ability to perform aerobic exercise
3. No current or recent (last 6 months) participation in a structured fitness program
4. Recent hospitalization for any reason (within the past three months)
5. Pregnant women
6. History of coronary artery disease, coronary bypass surgery or other cardiorespiratory events or conditions
7. Likely to experience clinically significant autonomic dysreflexia and/ or orthostatic hypotension in response to vigorous exercise
8. Any other conditions that the persons primary care physician deems is a contraindication to participation in arm ergometry exercise stress testing or vigorous exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Koontz, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HIIT: Exercise sessions will be 3x/week for 6 weeks (2 sessions supervised, 1 session unsupervised).
  HIIT: A handcycle or tabletop ergometer will be used for HIIT. Exercise sessions will be scheduled 3x/week for 6 weeks (2 sessions supervised, 1 session unsupervised). The HIIT goal is to achieve 10 sets of 60 second bouts of arm cycling at 90% of their PPO with 60 seconds of active recovery.
  Supervised exercise sessions: Measures include HR, BP, RPEs, Feeling Scale, and PPO. After warming up, individualized work/rest phases will be prescribed based on their PPO from their maximal aerobic test. Participants will be held at 90% PPO as a constant target intensity to start, shortening the work phase, and if necessary, lengthening the recovery phase. These parameters will be progressed each session. The trainer will determine when to change their work/rest parameters
Period: Overall Study
Arm/Group | HIIT
Started | 10
Completed | 7
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | HIIT
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Wrist Pain [Mean (Standard Deviation); unit: score on a scale] — Measured using the Numerical Rating Scale and averaged across sides (right and left). The scale ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
  score on a scale | 0.4 (0.97)
Elbow Pain [Mean (Standard Deviation); unit: score on a scale] — Measured using the Numerical Rating Scale and averaged across sides (right and left). The scale ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
  score on a scale | 0.6 (1.1)
Shoulder Pain [Mean (Standard Deviation); unit: score on a scale] — Measured using the Numerical Rating Scale and averaged across sides (right and left). The scale ranges from 0 (no pain) to 10 (pain as bad as you can imagine).
  score on a scale | 0.75 (1.5)
Shoulder Pain During Activity [Mean (Standard Deviation); unit: score on a scale] — Measured using the Wheelchair Users Shoulder Pain Index. The summative scale ranges from 0 to 150 with higher scores indicating higher levels of shoulder pain during activities of daily living.
  score on a scale | 8.5 (21.4)
General Health & Function [Mean (Standard Deviation); unit: score on a scale] — Scores generated on the Short Form 36 walk-wheel. Participants self report on health questions within 8 domains each of which are scored from 0 to 100. The scores from each of the subscales are then averaged together to obtain an overall total score. A score of 0 represents the worst possible health state and a score of 100 represents the best possible health state.
  score on a scale | 80.4 (12.6)
Physical Activity Status [Mean (Standard Deviation); unit: score on a scale] — Measured using the physical activity scale for individuals with physical disabilities (PASIPD). The higher the score the more active the individual (scores range from 0 to 199.5 metabolic equivalent hours/day).
  score on a scale | 24.8 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: HIIT Times
Description: Number of HIIT Work/Rest Times (number of intervals) completed by the participants per session (averaged over all sessions and participants)
Time Frame: To be recorded weekly, throughout study completion (3x/week for 6 weeks)
Population: Analysis performed only on the numbers of participants who completed at least one HIIT training session (n=9)
Measure: Mean (Standard Deviation); unit: Intervals
Groups:
- HIIT: Exercise sessions will be 3x/week for 6 weeks (2 sessions supervised, 1 session unsupervised).
  HIIT: A handcycle or tabletop ergometer will be used for HIIT. Exercise sessions will be scheduled 3x/week for 6 weeks (2 sessions supervised, 1 session unsupervised). The HIIT goal is to achieve 10 sets of 60 second bouts of arm cycling at 90% of their PPO with 60 seconds of active recovery.
  Supervised exercise sessions: Measures include HR, BP, RPEs, Feeling Scale, and PPO. After warming up, individualized work/rest phases will be prescribed based on their PPO from their maximal aerobic test. Participants will be held at 90% PPO as a constant target intensity to start, shortening the work phase, and if necessary, lengthening the recovery phase. These parameters will be progressed each session. The trainer will determine when to change their work/rest parameters based off of HR and RPEs.
  Unsupervised exercise sessions: Participants will repeat the same HIIT protocol they performed
Arm/Group | HIIT
Number analyzed (Participants) | 9
Intervals | 10 (0)

2. Primary Outcome: Power
Description: Change in peak power output (watts) pre and post HIIT training.
Time Frame: Baseline and 6 weeks
Population: The analysis was performed on the subset of subjects (n=6) who completed at least 12 supervised HIIT sessions and both the baseline and followup testing.
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | HIIT
Number analyzed (Participants) | 6
Watts | 5 (8.4)
Statistical Analysis 1: Comparison: HIIT; Test type: Superiority; p = .203, t-test, 2 sided

3. Primary Outcome: Cardiopulmonary Measures
Description: Change in Peak Oxygen Consumption (VO2) pre and post HIIT training (measured in mL/kg/min)
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | HIIT
Number analyzed (Participants) | 6
ml/kg/min | 0 (1.8)
Statistical Analysis 1: Comparison: HIIT; Test type: Superiority; p = 0.931, t-test, 2 sided

4. Primary Outcome: Cardiopulmonary Measures
Description: Peak heart rates achieved during each work interval within a training session were averaged together and then averaged over all training sessions and expressed as a percentage of the participant's maximum heart rate obtained at baseline, during training, or at the 6 week followup whichever value was highest. The peak training heart rates were then averaged across all participants to provide an overall measure of physical effort exerted by the group during HIIT exercise.
Time Frame: Recorded during each training session (3x/week for 6 weeks)
Population: Analysis performed only on the numbers of participants who completed at least one HIIT training session (n=9)
Measure: Mean (Standard Deviation); unit: percentage of maximum heart rate
Arm/Group | HIIT
Number analyzed (Participants) | 9
percentage of maximum heart rate | 94.1 (0.03)

5. Primary Outcome: Enjoyment of HIIT
Description: Measured using the Physical Activity Enjoyment Scale (PACES). The summative score ranges from 18 to 126 with higher scores indicating higher levels of enjoyment
Time Frame: 6 weeks
Population: Analysis performed only on the numbers of participants who completed at least one HIIT training session (n=9)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HIIT
Number analyzed (Participants) | 9
units on a scale | 114.8 (11.3)

6. Primary Outcome: Acceptability of HIIT
Description: Measured using the scores on one question on the Exercise Evaluation Form: "Rate your overall experience with the exercise intervention". Scores ranged from 5 (Very Satisfied) to 1 (Very Dissatisfied).
Time Frame: 6 weeks
Population: Analysis performed only on the numbers of participants who completed at least one HIIT training session (n=9)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIIT
Number analyzed (Participants) | 9
score on a scale | 5 (0)

7. Primary Outcome: Percentage of Participants Completing All Supervised Training Sessions
Description: The number of participants who completed all the supervised training sessions (12 sessions over 6 weeks) as a percentage of the total number of participants who completed the 6 week study. The HIIT program was considered feasible if a majority of participants (80% or more) were able to complete all 12 supervised training sessions in the 6 week study time frame.
Time Frame: To be recorded throughout study completion (6 weeks)
Population: Three participants were not included in the analysis because they had withdrawn from the study.
Measure: Number; unit: percent of participants
Arm/Group | HIIT
Number analyzed (Participants) | 7
percent of participants | 85.7

8. Secondary Outcome: Perceived Exertion
Description: The highest reported perceived exertion recorded during each HIIT exercise session was measured using the Borg Scale (6-20). The higher the number, the more perceived exertion felt during the activity. The perceived exertion ratings for all the sessions were averaged for each participant and then were averaged across all participants to provide an overall measure of perceived exertion felt by the group during HIIT exercise.
Time Frame: Recorded during each training session (3x/week for 6 weeks)
Population: Analysis performed only on the numbers of participants who completed at least one HIIT training session (n=9)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIIT
Number analyzed (Participants) | 9
score on a scale | 18.8 (1.4)

9. Secondary Outcome: Perceived Exertion (Adapted)
Description: Measured using the Wheel Scale (6-20)
Time Frame: To be recorded during each training session (3x/week for 6 weeks)
Population: This scale was found to be redundant and confusing to participants as the questions were similar to the Borg Scale but the score anchoring was different. It was not recorded for any participants.
Arm/Group | HIIT
Number analyzed (Participants) | 0

10. Secondary Outcome: Feelings During HIIT
Description: Lowest feeling score reported during the HIIT training and averaged across participants. The Feeling Scale score ranges from -5 (very bad) to +5 (very good).
Time Frame: Recorded during each training session (3x/week for 6 weeks)
Population: Analysis performed only on the numbers of participants who completed at least one HIIT training session (n=9)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HIIT
Number analyzed (Participants) | 9
units on a scale | -0.11 (2.8)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | HIIT
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIIT (N=10)
Pressure ulcer onset (Skin and subcutaneous tissue disorders) | 1 — Participant developed a pressure ulcer during the intervention period and was unrelated to the study.
Femur fracture from fall (Musculoskeletal and connective tissue disorders) | 1 — Participant fell and was hospitalized during the intervention period. The fall was unrelated to the the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT03152110/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT03152110/SAP_001.pdf